CLINICAL TRIAL: NCT02849002
Title: Non-Blinded Data Collection Study Of Concussion Using The BrainPulse
Brief Title: Un-blinded Data Collection Study of Concussion Using the BrainPulse(TM)
Status: Terminated | Type: Observational
Why Stopped: Study was stopped at site due to insufficient funding to continue
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JMC-1601-P01
Record Dates: First submitted 2016-07-25; First posted 2016-07-29 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Interventional Device: The BrainPulse is used on a patient's head to non-invasively detect, amplify and capture the brain motion caused by pulsatile blood flow from the cardiac cycle.
  The BrainPulse consists of a reusable headset that contains the accelerometers used to measure motion caused by pulsatile blood flow. The system is powered by rechargeable battery pack. The headset is placed on the subject's head and outputs data to a data collector that forwards the data to the computer. Each accelerometer has an attached tip that makes contact with the subject's head through hair. The headset also includes a photoplethysmograph (PPG) that simultaneously captures the subject's heart-rate information. There is no energy delivered to the brain or subject by these highly sensitive sensors.
  Interventions: Device: BrainPulse

INTERVENTIONS:
Device: BrainPulse — Jan Medical's BrainPulse measures the brain motion caused by pulsatile blood flow from the cardiac cycle, referred to as the BrainPulse signal. The BrainPulse measures skull acceleration in response to the brain motion using an array of sensors placed on the head.
  Other Names: BrainPulse 1100

SUMMARY:
The primary objective of this study is to collect un-blinded BrainPulse recordings from youth and adults that have a confirmed diagnosis of concussion per protocol guidelines in order to improve a concussion detection algorithm previously developed by Jan Medical, Inc. Subjects will be followed for 21 days after the initial injury with BrainPulse recordings to study the subject's recovery process. The symptomatic evaluation, physical examination, and BrainPulse recordings will be entered in a database to assess clinical outcome and device utilization.BrainPulse(TM)

DETAILED DESCRIPTION:
Jan Medical is conducting a data collection study with the goal of developing further insight into understanding the signal features within a BrainPulse recording that are only present when the subject has a confirmed concussion. The initial pilot blinded study with Stanford University showed that there is increased energy in the 8-15 Hz range for BrainPulse recordings from adolescent male football players with a confirmed concussion. The current un-blinded study is designed to record the BrainPulse signal from a more diverse subject population to represent patients who have been diagnosed with a concussion in clinic setting. Subjects will include males and females ages 13 and older.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 13 years old and not part of any other vulnerable population such as pregnant women.
2. Suspected or confirmed concussion by medical professional
3. Not more than 3 days since injury/trauma event
4. Willing and able to participate in all required study evaluations and allow access to medical testing and records
5. Signed informed consent/assent, and/or have a legally authorized representative willing to provide informed consent on behalf of the subject.
6. Demonstrates a minimum of 3 of the following symptoms:

   * Headache
   * Pressure in head
   * Dizziness
   * Neck pain
   * Fatigue/ low energy
   * Nausea or vomiting
   * Irritability
   * Difficulty in concentrating/performing tasks
   * Memory impairment
   * Insomnia
   * Reduced tolerance to stress
   * Sensitivity to light
   * Difficulty balancing
   * Blurred vision
   * Confusion
   * More emotional than usual
   * Sadness
   * Nervous/Anxious
   * Vacant stare
   * Delayed verbal/motor response
   * 'Feeling like in a fog'
   * 'Don't feel right'

Exclusion Criteria:

1. Wound or open laceration on the head in the area of one of the BrainPulse sensors that would impede use of the BrainPulse device
2. Any serious medical condition that in the opinion of the medical professional would impair ability to provide informed consent/assent or otherwise disqualify a patient from participation
3. Currently participating in or planning to participate in another clinical study during the course of the current clinical study.
4. Implantation of any medical device in head (e.g. ventriculoperitoneal shunt)
5. An alternative diagnosis is made other than concussion

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults, ages 13 and older, who are diagnosed with a concussion or mild Traumatic Brain Injury (mTBI), typically due to a trauma event such as a fall, sports injury, motor vehicle accident, etc.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
Number of BrainPulse recordings from suspected and confirmed concussed subjects | Through study completion, expected to be 6 months
  collect un-blinded BrainPulse recordings from youth and adults that have a confirmed diagnosis of concussion per protocol guidelines in order to improve a concussion detection algorithm previously developed by Jan Medical, Inc.The primary endpoint is to enroll and record BrainPulse signals from 500 subjects with a suspected concussion. To gather sufficiently diverse data, at least 300 participants will have had a confirmed diagnosis of concussion. The data will be used to improve the algorithm for aiding in the diagnosis of concussion.

SECONDARY OUTCOMES:
Average number of days the signal pattern seen within BrainPulse recordings from confirmed concussed subjects from the initial recording persist over the course of the 21 day follow up period. | Through study completion, expected to be 1 year]
  The secondary endpoint is to assess the differences in BrainPulse recordings between the initial visit and each subsequent follow-up visit to better understand the recovery process post concussion.

CONTACTS AND LOCATIONS:
Overall Officials: Neilank Jha, MD, Principal Investigator — Konkussion
Locations (1):
- Konkussion Inc., Woodbridge, Ontario, Canada